CLINICAL TRIAL: NCT03254355
Title: Efficacy of Physiotherapy for Urinary Incontinence in Women With a Known Avulsion Injury of the Puborectalis Muscle: A Randomized Controlled Trial
Brief Title: Efficacy of Physiotherapy for Urinary Incontinence in Women With a Puborectalis Avulsion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Mélanie Morin, Researcher and Associate Professor, Université de Sherbrooke
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MP-31-2018-1758
Record Dates: First submitted 2017-08-09; First posted 2017-08-18 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Urinary Incontinence; Postpartum; Pelvic Floor; Perineal Rupture, Obstetric; Physiotherapy
Keywords: avulsion injury; urinary incontinence; multimodal physiotherapy
MeSH Terms: conditions — Urinary Incontinence; Fractures, Avulsion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multimodal physiotherapy (Experimental): 12 weeks of weekly multimodal physiotherapy treatments
  Interventions: Procedure: Multimodal physiotherapy
- Waiting-list control group (No Intervention): 12 weeks of weekly full-body relaxation massage

INTERVENTIONS:
Procedure: Multimodal physiotherapy — 12 weeks of weekly physiotherapy treatments including education segment, electrical stimulation and PFM exercises consisting of strength, endurance and coordination exercises accompanied by biofeedback
  Arms: Multimodal physiotherapy

SUMMARY:
Childbirth is a major risk factor for pelvic floor muscle (PFM) trauma. In one third of women, stretching of the PFM will result in an avulsion injury (i.e. disconnection of the muscle from its insertion points on the pubic symphysis). Recent advances in imaging have led to the discovery of this previously unknown major injury and further research now enables its diagnosis with readily available techniques. Avulsion injury has alarming consequences because it has been associated with a higher rate of urinary incontinence in the postpartum period as well as the long-term development of other major urogynecological conditions such as pelvic organ prolapse and anal incontinence. Women with avulsion not only suffer from severe symptoms with significant related impacts on physical activities, overall well-being and quality of life, but they also present a higher rate of surgical failures. Moreover, it is still unknown whether the most recommended first-line treatment for urinary incontinence -PFM physiotherapy- is effective in women with this major trauma. Until now, only a pilot study conducted by our team supports the rationale and the efficacy of physiotherapy for improving PFM function in women with avulsion, despite their major muscle injury.

Primary objective: To evaluate the efficacy of physiotherapy for urinary incontinence in women with avulsion at 9-months after randomization compared to a waiting-list control group.

Secondary objectives:

1. To compare physiotherapy to the control group after treatment and at 9-months after randomization in terms of: a) incontinence and prolapse (objective quantification, symptoms and related impact); b) PFM morphology and function; c) sexual function; d) self-efficacy; e) cost analysis; f) treatment satisfaction and impression of change.
2. To investigate the impact of the severity of the avulsion (i.e. unilateral or bilateral) on the response to physiotherapy treatment on the aforementioned outcomes.

DETAILED DESCRIPTION:
This is a multicenter randomized controlled trial using a parallel group design that involves women with a confirmed diagnosis of avulsion and suffering from urinary incontinence. Participants will be randomized into either physiotherapy or a waiting-list control group. Both groups will be evaluated at baseline, post-treatment (3 months post-randomization) and 9 months after randomization. Women in the control group will receive full-body relaxation massage which has shown no effect on continence but was selected to control for effects of attention received by the therapist. After the 9-month assessment, women assigned to the control group will receive the same physiotherapy treatment and undergo a last assessment.

ELIGIBILITY:
Inclusion Criteria:

* 18-45 years old
* Postpartum women (≥ 1 vaginal delivery at term (≥ 37 weeks) and ≥ 3 months postpartum
* ≥ 3 urinary incontinence episodes per week over the last 3 months (Symptoms of incontinence must be associated predominantly or solely with stress urinary incontinence (as opposed to urge incontinence) which will be determined with a recommended and validated diagnosis questionnaire (Questionnaire for Urinary Incontinence Diagnosis))
* Women with diagnosis avulsion injury

Exclusion Criteria:

* Pregnancy or postmenopausal
* Previous pelvic irradiation, urogynecological surgery, or PFM physiotherapy after the avulsion occurred
* Significant prolapse (≥3 degree)
* Incontinence due to other causes such as infection, neurological diseases, voiding difficulties
* Any other acute or chronic medical problems likely to interfere with treatment or evaluation such as cancer, chronic constipation (Rome III criteria), obesity (body mass index >35), pacemaker, bladder stimulator
* Medication or ongoing treatment likely to interfere with incontinence

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 126 (Actual)
Dates: Start 2017-08-28 (Actual); Primary Completion 2023-05-10 (Actual); Study Completion 2023-05-10 (Actual)

PRIMARY OUTCOMES:
Percent reduction in the number of urinary incontinence episodes | baseline, post-treatment (3 months post-randomization) and 9 months after randomization
  The 7-day bladder diary was selected as the primary outcome to measure urinary leakage reduction

SECONDARY OUTCOMES:
Change in symptoms and impact of incontinence and other urogynecological conditions | baseline, post-treatment (3 months post-randomization) and 9 months after randomization
  Evaluated with ICI Modular Questionnaires (ICIQ), Pelvic Floor Distress Inventory (PFDI), Pelvic Floor Impact Questionnaire (PFIQ-SF) and Pelvic Organ Prolapse Symptom score (POP-SS)
Change in pelvic floor muscle morphometry and function | baseline, post-treatment (3 months post-randomization) and 9 months after randomization
  Evaluated with transperineal ultrasound and dynamometry
Change in severity of prolapse | baseline, post-treatment (3 months post-randomization) and 9 months after randomization
  Evaluated with POP-Q assessment
Change in sexual function | baseline, post-treatment (3 months post-randomization) and 9 months after randomization
  Evaluated with Female Sexual Function Index (FSFI) and Pelvic Organ Prolapse/Incontinence Sexual Questionnaire (PISQ-SF)
Change in self-efficacy | baseline, post-treatment (3 months post-randomization) and 9 months after randomization
  Evaluated with Broom Pelvic Muscle Self-Efficacy Scale
Cost analysis | baseline and 9 months after randomization
  Evaluated with Dowell-Bryant Incontinence Cost Index (DBICI)
Treatment satisfaction and impression of change | baseline, post-treatment (3 months post-randomization) and 9 months after randomization
  Evaluated with Patient Satisfaction Questionnaire (PSQ) and Patient's Global Impression of Change (PGIC)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec, Canada